CLINICAL TRIAL: NCT04654091
Title: Cryotherapy With Liquid Nitrogen and Nitric-zinc Complex in the Treatment of Plantar Warts. Randomised Controlled Trial.
Brief Title: Cryotherapy VS. Nitric-zinc Complex in the Treatment of Plantar Warts.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Sara García Oreja, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/471-R_X_TesisUCM
Record Dates: First submitted 2020-11-22; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Plantar Wart
Keywords: plantar wart; nitric acid; cryotherapy

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoteraphy with liquid nitrogen (Experimental): Patients older than 18 years with a diagnosis of plantar wart, who have agreed to participate in the study.
  Interventions: Procedure: Cryoteraphy with liquid nitrogen
- Nitric-zinc complex (Experimental): Patients older than 18 years with a diagnosis of plantar wart, who have agreed to participate in the study.
  Interventions: Procedure: Nitric-zinc complex

INTERVENTIONS:
Procedure: Cryoteraphy with liquid nitrogen — Weekly, at each visit, before applying the treatment, a debridement of the hyperkeratotic tissue covering the wart will be performed with a scalpel handle of number 3 and a scalpel blade of number 15, and then the treatment will be applied.
  Subsequently, the application of cryotherapy with liquid nitrogen will be carried out using CryoPen b® (HO Equipment, Hhislenghien-Belgium). To analyze the homogeneous application in all the patients in the study, perform 2 applications of 15 seconds per session, with an interval of 30 seconds between each application, such and as manufacturers recommend. The number of sessions in which the product is applied will be a maximum of 5, following the procedure of previous studies.
  Arms: Cryoteraphy with liquid nitrogen
Procedure: Nitric-zinc complex — Weekly, at each visit, before applying the treatment, a debridement of the hyperkeratotic tissue covering the wart will be performed with a scalpel handle of number 3 and a scalpel blade of number 15, and then the treatment will be applied.
  Subsequently, the application of nitric acid-zinc complex with Verrutop® (Isdin, Barcelona-Spain) will be carried out. The preparation is applied by making small touches with the applicators included in the product.
  The number of sessions in which the product is applied will be a maximum of 5, following the recommendations of the manufacturers in the product data sheet.
  Arms: Nitric-zinc complex

SUMMARY:
Plantar warts are benign skin lesions caused by human papillomavirus (HPV).There are several treatment methods for this illness, but none of them can heal all patients. Cryotherapy using liquid nitrogen is one of the most common local treatments. In this study, we will compare the effectiveness of cryotherapy with liquid nitrogen with the association of organic acids and nitric acid (nitric-zinc complex). In addition, as secondary objectives have been defined: 1) know the number of applications necessary for each treatment to achieve the complete resolution of the plantar wart, in order to compare the healing times between each treatment and establish which treatment is faster, 2) analyze the influence of the HPV biotype, the location of the lesion and the time of evolution in the response to the different treatments, and 3) Compare the ultrasound signs of plantar warts with the ultrasound signs of healthy skin after the resolution of the process.

DETAILED DESCRIPTION:
A randomized controlled clinical trial is proposed. The recruitment of patients will be carried out by including the sample of those patients who have diagnostic confirmation of plantar wart in the Chiropodology and Surgery Service of the University Podiatry Clinic of the Complutense University of Madrid, consecutively, between November 2020 and the date when the estimated sample size is reached.

Participants in the trial will be assigned with equal probability to each treatment arm, based on their consecutive inclusion in the study. Subsequently, the treatment allocation will be determined by a random code generated by the Epidat 4.1 program using random permuted blocks. The treatment used will be evident both for the participant and for the research podiatrist responsible for the intervention. However, the primary result will be confirmed by the microbiological study carried out by the Department of Microbiology of the Complutense University of Madrid, which does not know any data about the patient or the treatment group to which it was initially assigned.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 12 years.
* Patients diagnosed with recalcitrant or non-recalcitrant plantar wart.

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus.
* Peripheral vascular disease.
* Patients with an immune system disorder or in immunosuppressants treatment.
* Peripheral or central neuropathy.
* Coagulation disorders.
* Raynaud's disease or some alteration of the perception of cold or heat.
* Alterations in healing for wounds or in the synthesis of collagen.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cryotherapy efficacy versus nitric-zinc complex | One year approximately
  Compare the cure rates of the following topical treatments of plantar warts: cryotherapy with liquid nitrogen; and the association of organic acids and nitric acid (nitric-zinc complex), in a period of 12 weeks.
  A polymerase chain reaction (PCR) test will be performed when there is an absence of clinical signs and symptoms of plantar wart, considering cure when a negative result is obtained.
  In those patients in whom the maximum number of treatment sessions recommended in the technical sheet of each product has been carried out and clinical signs of plantar wart are still observed, as well as in those patients who after 12 weeks of follow-up continue to present signs and symptoms Clinicians will be considered as not cured, considering the study ended.

SECONDARY OUTCOMES:
Number of applications | One year approximately
  Know the number of applications needed for each treatment to achieve full resolution of the plantar wart, a fin to compare the healing times between each treatment and establish which treatment is faster.
Influence of the characteristics of the lesion | One year approximately
  To analyze the influence of the HPV biotype, the location of the lesion and the time of evolution in the response to the different treatments.
Ultrasound signs of plantar warts | One year approximately
  Compare the ultrasound signs of plantar warts with the ultrasound signs of healthy skin after the resolution of the process.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Álvaro Afonso, PhD, Principal Investigator — Universidad Complutense de Madrid